CLINICAL TRIAL: NCT05104749
Title: Homeopathic Treatment of Post-acute COVID-19 Syndrome- A Pilot Randomized Controlled Trial
Brief Title: Homeopathic Treatment of Post-acute COVID-19 Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Southwest College of Naturopathic Medicine (Other)
Collaborators: Samueli Institute for Information Biology (Other)
Responsible Party: Principal Investigator, Elizabeth Rice, Associate Professor Interim Dept Chair Homeopathy and Pharmacology, Southwest College of Naturopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0012021
Record Dates: First submitted 2021-10-28; First posted 2021-11-03 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Post-acute Covid-19 Syndrome
Keywords: Long Covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both study medication and placebo are identical in appearance, odor, and taste. Statistician will be blinded as to treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Homeopathic Treatment Group (Experimental): Individualized homeopathic medicines on impregnated lactose pellets will be prescribed to each participant based on the totality of their physical, emotional, and mental symptoms. All medicines prescribed are listed in the Homeopathic Pharmacopoeia of the United States (HPUS) as outlined in the Food, Drug, and Cosmetics Act of 1939
  Interventions: Drug: Homeopathic Medication
- Placebo Group (Placebo Comparator): Identical lactose pellets in size, odor, and taste without the impregnated homeopathic medicines.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Homeopathic Medication — Homeopathic medicines are prepared according to standardized methods as specified by the Homeopathic Pharmacopoeia of the United States (HPUS), which was mandated by Congress to regulate the manufacture of homeopathic medicines as part of the Food, Drug, and Cosmetics Act of 1939. All homeopathic medicines prescribed in this study must be found in the HPUS. For a complete list of homeopathic medicines, contact the researchers.
  Arms: Homeopathic Treatment Group
Other: Placebo — Inert lactose pellets
  Arms: Placebo Group

SUMMARY:
To determine whether an individually prescribed homeopathic medicine has an effect greater than a placebo and is a viable treatment option to improve fatigue and quality of life for patients suffering from the symptoms of Post-acute COVID-19 Syndrome. The researchers hope to achieve this goal by conducting a clinical trial that is scientifically rigorous and clinically relevant. Expected results of this pilot study will be to obtain sufficient experience and preliminary feasibility data to justify a larger clinical trial of this hypothesis.

DETAILED DESCRIPTION:
The researchers objectives for the study are to: 1) identify efficient means of recruiting subjects, 2) test and refine the initial study design and treatment protocol, 3) evaluate the instruments for assessing treatment outcomes, 4) estimate sample sizes that will be required in the full-scale trial, 5) determine which homeopathic medicines are most often prescribed for this syndrome, and 6) determine whether there is a measurable effect size difference or positive trend in reduction of symptoms in patients treated with homeopathy.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-64
* Any ethnicity
* Adequate cognitive function to be able to give informed consent
* Technologically competent to complete web forms and perform video calls
* Positive PCR test (polymerase chain reaction) result for SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2)
* Persistent fatigue for a minimum of 60 days since diagnosis of Covid-19.
* A fatigue score above 21 in the Fatigue Assessment Scale upon enrollment
* Willing to fill out regular questionnaires
* Willing to use homeopathic medicines

Exclusion Criteria:

* Clinically significant kidney, heart, or hepatic impairment as determined by clinical judgment

  * Previous hospitalization in ICU for Covid-19
  * Diagnosis of Chronic Fatigue Syndrome, Fibromyalgia, or Lyme disease prior to Covid-19
  * Chronic psychiatric illness or neurological illness prior to Covid-19 diagnosis Taking opioid analgesics, opioid dependence or undergoing treatment for substance abuse or addiction
  * Taking steroid medication or immunosuppressive medications
  * Suspected or confirmed pregnancy or breastfeeding
  * Active cancers
  * Current treatment by a homeopathic practitioner
  * Initiation of another treatment for Long Covid within the past 2 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Rice, ND, Principal Investigator — Southwest College of Naturopathic Medicine
Locations (1):
- Southwest College of Naturopathic Medicine, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Homeopathic Treatment Group: Long Covid patients received individualized homeopathic treatment with homeopathic medicines. Dosage and frequency of administration was determined by each provider on an individualized basis.
- Placebo Group: Long Covid patients received placebo homeopathic medicines (i.e. identical lactose pellets in size, odor, and taste without the impregnated homeopathic medicines)
Period: Overall Study
Arm/Group | Homeopathic Treatment Group | Placebo Group
Started | 38 | 39
Completed | 36 | 36
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Population: All participants under randomization were included (intention-to-treat population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Homeopathic Treatment Group | Placebo Group | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (8.3) | 44.4 (11.1) | 42.9 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 38 | 72
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 34 | 35 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Education Status [Count of Participants; unit: Participants]
  High School | 0 | 1 | 1
  Some college | 12 | 16 | 28
  Bachelor's Degree | 17 | 12 | 29
  Master's Degree | 8 | 9 | 17
  PhD or higher | 1 | 1 | 2
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.6 (7.8) | 26.2 (4.8) | 26.9 (6.5)
Duration of Long Covid Symptoms [Mean (Standard Deviation); unit: Days] | 246.4 (141.0) | 285.5 (151.1) | 266.2 (146.6)
Hospitalization Rate for Acute Covid-19 Infection [Count of Participants; unit: Participants] — At baseline, all participating subjects receiving placebo or homeopathy were assessed for hospitalization during their initial COVID-19 acute infection.
  Participants | 3 | 6 | 9
Number of Vaccinated Participants [Count of Participants; unit: Participants] — At baseline, all participating subjects receiving placebo or homeopathy were assessed whether they had received a full or partial COVID-19 vaccination.
  Participants | 29 | 30 | 59
Number of Long Covid Booster Participants [Count of Participants; unit: Participants] — At baseline, all participating subjects receiving placebo or homeopathy were assessed whether they had received a COVID-19 booster vaccination.
  Participants | 11 | 14 | 25
Number of Medications [Count of Participants; unit: Participants]
  Zero | 15 | 15 | 30
  1-2 | 10 | 12 | 22
  3 or more | 13 | 12 | 25
Number of Supplements [Count of Participants; unit: Participants]
  Zero | 5 | 11 | 16
  1-4 | 17 | 14 | 31
  5 or more | 16 | 14 | 30
Baseline Score in Fatigue Assessment Scale [Mean (Standard Deviation); unit: score on a scale] — The Fatigue Assessment Scale (FAS) is a 10-item self-report scale evaluating symptoms of chronic fatigue. The total score ranges from 10 to 50, with a higher score indicating more severe fatigue.
  Less than 22 indicates "normal" (i.e. healthy) levels of fatigue between 22 and 34 indicates mild-to-moderate fatigue 35 or more indicates severe fatigue (Hendricks et al., 2018).
  score on a scale | 34.4 (7.1) | 35.8 (6.8) | 35.1 (7.0)
Baseline Score in SF-36 Physical Composite Score (PCS) [Mean (Standard Deviation); unit: score on a scale] — Quality of life was evaluated by using the the RAND 36-Item Short Form Health Survey (SF-36), which was completed by participants throughout the study. The SF-36 evaluates 8 health concepts and can be aggregated into two summary scores: the Physical (PCS) and Mental (MCS) Component Summary scores.
  Each item of the scale ranges from 0-100, where high values mean good health status, while lower values indicate poor health status. Items are averaged together to create PCS or MCS scale scores.
  score on a scale | 45.8 (17.4) | 42.9 (20.4) | 44.3 (18.9)
Baseline Score in SF-36 Mental Combined score (MCS) [Mean (Standard Deviation); unit: score on a scale] — Quality of life was evaluated by using the the RAND 36-Item Short Form Health Survey (SF-36), which was completed by participants throughout the study. The SF-36 evaluates 8 health concepts and can be aggregated into two summary scores: the Physical (PCS) and Mental (MCS) Component Summary scores.
  Each item of the scale ranges from 0-100, where high values mean good health status, while lower values indicate poor health status. Items are averaged together to create PCS or MCS scale scores.
  score on a scale | 35.7 (18.3) | 37.6 (16.7) | 36.6 (17.4)
Baseline Score in PHQ-9 [Mean (Standard Deviation); unit: score on a scale] — The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool for assessing depression The PHQ-9 scores each of the 9 DSM-IV depression criteria as "0" (not at all) to "3" (nearly every day).
  PHQ-9 scores range from 0 to 27, with scores of 5, 10, 15, and 20 representing mild, moderate, moderately severe, and severe depression, respectively
  score on a scale | 12.8 (5.6) | 10.8 (5.1) | 11.8 (5.4)
Baseline Score in MYMOP Symptom #1 [Mean (Standard Deviation); unit: score on a scale] — The Measure Yourself Medical Outcomes Profile (MYMOP) is a problem specific and individualized measure that captures what patients consider are the two most important symptoms associated with their condition (Long COVID) and an activity of daily living that is affected by these symptoms.
  The symptom is then rated by the patient on a scale 0-6 where higher values mean poor health and lower values indicate good health.
  score on a scale | 4.6 (1.2) | 4.5 (1.0) | 4.5 (1.1)
Baseline Score in MYMOP Symptom #2 [Mean (Standard Deviation); unit: score on a scale] — The Measure Yourself Medical Outcomes Profile (MYMOP) is a problem specific and individualized measure that captures what patients consider are the two most important symptoms associated with their condition (Long COVID) and an activity of daily living that is affected by these symptoms.
  The symptom is then rated by the patient on a scale 0-6 where higher values mean poor health and lower values indicate good health.
  score on a scale | 4.4 (1.0) | 4.4 (1.0) | 4.4 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Assessment Scale (FAS)
Description: The Fatigue Assessment Scale (FAS) is a 10-item self-report scale evaluating symptoms of chronic fatigue. The total score ranges from 10 to 50, with a higher score indicating more severe fatigue. Less than 22 indicates "normal" (i.e. healthy) levels of fatigue between 22 and 34 indicates mild-to-moderate fatigue 35 or more indicates severe fatigue (Hendricks et al., 2018).
Time Frame: Baseline, 4, 8 and 12 weeks
Population: All patients under randomization were included (intention-to-treat population) regardless whether or not they adhered to the treatment protocol or provided complete data sets.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Homeopathic Treatment Group | Placebo Group
Number analyzed (Participants) | 36 | 36
score on a scale
  4 Weeks | 32.9 (7.6) | 31.4 (7.7)
  8 Weeks | 29.0 (8.0) | 27.4 (9.4)
  12 Weeks | 29.4 (9.1) | 27.3 (10.0)

2. Primary Outcome: SF-36 Physical Composite Score (PCS)
Description: Quality of life was evaluated by using the the RAND 36-Item Short Form Health Survey (SF-36), which was completed by participants throughout the study. The SF-36 evaluates 8 health concepts and can be aggregated into two summary scores: the Physical (PCS) and Mental (MCS) Component Summary scores.
  Each item of the scale ranges from 0-100, where high values mean good health status, while lower values indicate poor health status. Items are averaged together to create PCS or MCS scale scores.
Time Frame: Baseline and 4, 8, and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Homeopathic Treatment Group | Placebo Group
Number analyzed (Participants) | 36 | 36
score on a scale
  4 Weeks | 51.8 (18.2) | 51.1 (22.3)
  8 Weeks | 55.0 (22.6) | 58.7 (26.5)
  12 Weeks | 55.0 (23.1) | 61.2 (27.4)

3. Primary Outcome: SF-36 Mental Composite Score (MCS)
Description: Quality of life was evaluated by using the the RAND 36-Item Short Form Health Survey (SF-36), which was completed by participants throughout the study. The SF-36 evaluates 8 health concepts and can be aggregated into two summary scores: the Physical (PCS) and Mental (MCS) Component Summary scores.
  Each item of the scale ranges from 0-100, where high values mean good health status, while lower values indicate poor health status. Items are averaged together to create PCS or MCS scale scores.
  ￼
Time Frame: Baseline and 4, 8, and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Homeopathic Treatment Group | Placebo Group
Number analyzed (Participants) | 36 | 36
score on a scale
  Week 4 | 43.0 (21.6) | 50.2 (21.7)
  Week 8 | 47.8 (22.0) | 54.7 (24.8)
  Week 12 | 49.8 (23.4) | 57.3 (25.7)

4. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9)
Description: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool for assessing depression The PHQ-9 scores each of the 9 DSM-IV depression criteria as "0" (not at all) to "3" (nearly every day).
  PHQ-9 scores range from 0 to 27, with scores of 5, 10, 15, and 20 representing mild, moderate, moderately severe, and severe depression, respectively.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Homeopathic Treatment Group | Placebo Group
Number analyzed (Participants) | 36 | 36
score on a scale | 7.8 (5.7) | 6.8 (4.8)

5. Secondary Outcome: Measure Yourself Medical Outcomes Profile Symptom #1
Description: The Measure Yourself Medical Outcomes Profile (MYMOP) is a problem specific and individualized measure that captures what patients consider are the two most important symptoms associated with their condition (Long COVID) and an activity of daily living that is affected by these symptoms.
  The symptom is then rated by the patient on a scale 0-6 where higher values mean poor health and lower values indicate good health.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Homeopathic Treatment Group | Placebo Group
Number analyzed (Participants) | 36 | 36
score on a scale | 1.3 (1.9) | 1.6 (1.8)

6. Secondary Outcome: Measure Yourself Medical Outcomes Profile Symptom #2
Description: as for outcome 5
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Homeopathic Treatment Group | Placebo Group
Number analyzed (Participants) | 36 | 36
score on a scale | 1.0 (1.7) | 1.7 (1.6)

7. Secondary Outcome: Patient Doctor Depth of Relationship (PDDR)
Description: The Patient Doctor Depth of Relationship (PDDR) scale is an eight item, patient self-completed questionnaire designed to measure patient-doctor relational depth. A single overall depth-of-relationship score can be calculated, which ranges from 0 (no relationship) to 32 (very strong relationship).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Homeopathic Treatment Group | Placebo Group
Number analyzed (Participants) | 36 | 36
score on a scale | 24.1 (6.4) | 24.3 (6.1)

ADVERSE EVENTS:
Time Frame: During study duration (12 weeks).
Arm/Group | Homeopathic Treatment Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/38 | 2/39
Other Adverse Events (participants affected / at risk) | 6/38 | 6/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Homeopathic Treatment Group (N=38) | Placebo Group (N=39)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) — Elevated blood pressure reading responded to cardiologist change in medication.
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Homeopathic Treatment Group (N=38) | Placebo Group (N=39)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
Vaccine Injury (Immune system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT05104749/Prot_SAP_000.pdf